CLINICAL TRIAL: NCT02685917
Title: Effects of Microfracture With/Without Collagen Augmentation in Patients Undergoing High Tibial Osteotomy: A Randomized, Controlled, Double-Blind Trial
Brief Title: Microfracture With/Without Collagen Augmentation in Patients Undergoing High Tibial Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Collagen augmentation
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Collagen Augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microfracture with Collagen Augmentation in HTO (Experimental): Two groups, either collagen augmentation or not. Firstly, all patients underwent an arthroscopic examination and microfracture for bone marrow. Collagen augmentation included Cartifill insertion after arthroscopic microfracture.
  Interventions: Procedure: Microfracture with Collagen Augmentation
- Microfracture without Collagen Augmentation in HTO (Active Comparator): Two groups, either collagen augmentation or not. Firstly, all patients underwent an arthroscopic examination and microfracture for bone marrow. Collagen augmentation included Cartifill insertion after arthroscopic microfracture.
  Interventions: Procedure: Microfracture without Collagen Augmentation

INTERVENTIONS:
Procedure: Microfracture without Collagen Augmentation — Cartifill applied for collagen augmentation
  Arms: Microfracture without Collagen Augmentation in HTO
Procedure: Microfracture with Collagen Augmentation — Cartifill applied for collagen augmentation
  Arms: Microfracture with Collagen Augmentation in HTO

SUMMARY:
The quality of cartilage regeneration after marrow stimulation is well documented to be unpredictable, because they do not regenerate consistent amount of cartilage. To overcome the shortcomings of the microfracture technique, various augmentation techniques using synthetic collagen matrix, scaffolds or plug devices have been developed. However, their efficacy remains unclear. The purpose of this prospective randomized controlled study is to evaluate whether the microfracture in combination with collagen gel augmentation could improve the quality of cartilage regeneration in patients undergoing medial open wedge high tibial osteotomy (HTO) for the treatment of medial unicompartmental knee osteoarthritis (OA).

DETAILED DESCRIPTION:
CartiFill™ (atelocollagen, Sewon Cellontech, Seoul, Korea) was developed to to provide a matrix stability and to maintain the blood clot in the defect site, which promoted the cartilage regeneration by mesenchymal stem cell . It was a atelocollagen, highly purified porcine derived type collagen І that has been modified to virtually eliminate the risk of rejection by removal of telopeptide.

The investigators randomized patients undergoing HTO in combination with microfracture to receive either microfracture alone (control group, n = 5) or microfracture with collagen augmentation (experimental group, n=6). At postoperative one year, the clinical outcome in terms of Visual Analogue Scale of pain level (VAS), Knee Injury and Osteoarthritis Outcome Score (KOOS), International Knee Documentation Committee (IKDC) score, and Tegner scores were evaluated. In addition, second look arthroscopic examination and biopsy of regenerated cartilage were carried out when the HTO plate was removed at postoperative one year. Biopsy specimens were graded by International Cartilage Repair Society Visual Assessment Scale (ICRS II scores). Finally, radiologic outcome in terms of Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scores was assessed using follow up MRI undertaken at postoperative one year.

ELIGIBILITY:
Inclusion Criteria:

* Aged below 65 years with isolated medial compartment osteoarthritis
* Good range of motion
* No ligament instability
* Having medicare insurance

Exclusion Criteria:

* Diagnosis of severe tricompartment osteoarthritis indicated for total knee arthroplasty
* Inflammatory arthritis(rheumatoid arthritis), osteonecrosis
* Flexion contracture ≥ 15°
* Knee range of motion < 120°
* Joint instability
* A history of knee joint infection and who refused to participate

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from Baseline score to score of postoperative 1 year.
International Knee Documentation Committee (IKDC) score | Change from Baseline score to score of postoperative 1 year.
Tegner score | Change from Baseline score to score of postoperative 1 year.

SECONDARY OUTCOMES:
The MRI observation of cartilage repair tissue (MOCART) score | Preoperative & postoperative 1 year.
International Cartilage Repair Society (ICRS) II scoring system | Postoperative 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — the Catholic Univerisity of Korea Seoul St Mary's hospital